CLINICAL TRIAL: NCT04917484
Title: Dosimetry Based PRRT Versus Standard Dose PRRT With Lu-177-DOTATOC in NEN Patients- a Randomized Study; a Step Towards Tailored PRRT
Brief Title: Dosimetry Based PRRT Versus Standard Dose PRRT With Lu-177-DOTATOC in NEN Patients
Acronym: DOBATOC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tine Gregersen, MD (Other)
Responsible Party: Sponsor-Investigator, Tine Gregersen, MD, Primary investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2019-002450-23
Record Dates: First submitted 2020-09-01; First posted 2021-06-08 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Neoplasm
Keywords: Peptide receptor radionuclide therapy; Dosimetry
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: Randomized, non blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): Patients in this arm receive our standard treatment. Four treatment with standard dose of 7.4 GBq Lu-177-DOTATOC
  Interventions: Drug: Lu-177-DOTA-Octreotide
- Dosimetry (Experimental): Patients in this treatment arm receive individualized calcuted treatment depending on kidney function and kidney dose. The treatment activity can differ from one treatment to the next.
  Interventions: Drug: Lu-177-DOTA-Octreotide

INTERVENTIONS:
Drug: Lu-177-DOTA-Octreotide — Lu-177-DOTATOC in standard doses or individualized doses.

SUMMARY:
In this study, we want to randomize patients with neuroendocrine neoplasms (NENs) who are eligible for peptide receptor radionuclide therapy (PRRT), to either standard PRRT consisting of 4 treatments with 7.4 GBq Lu-177-DOTATOC (standard arm) or 4 treatments with individualized doses of Lu-177-DOTATOC (dosimetry arm). In the dosimetry arm, the first dose depends on the patients' kidney function and thereafter the absorbed dose to the kidneys at the previous treatment. A max of 20GBq will be administered at the first treatment and 25GBq at treatment 2-4. We aim to reach an accumulated kidney dose of 24Gy.

After the first treatment all patients will go through three SPECT/CT scans 24 hours, 4 days, and 7 days, after treatment to calculate absorbed kidney dose. The patients in the standard dose treatment arm will have one SPECT/CT scan after each of the last three treatments; all performed 24 hours after treatment, used to approximate the kidney dose assuming the clearance of the Lu-177 DOTATOC is the same after all treatments. The patients in the dosimetry based treatment arm will go through three SPECT/CT scans after all four treatments for dosimetry calculation.

Bone marrow dosimetry is calculated after all treatments in the dosimetry based treatment arm and after the first treatment in the standard treatment arm. For bone marrow dosimetry, blood samples are drawn right before administration of Lu-177 DOTATOC (time 0) and 3 minutes, 45 minutes, 2 hours, 4 hours, 7-8 hours, 24 hours, 4 days, and 7 days after administration of Lu-177 DOTATOC.

Standard blood samples are routinely drawn every 2nd week after every treatment in all included patients and analysed regarding liver, kidney and bone marrow function. Kidney clearance is evaluated with Tc-DTPA clearance at baseline.

Blood and urinary samples will be collected at baseline and 3 months after the last treatment for kidney fibrosis analyses.

At baseline, blood and urine samples are collected for a biobank. All included patients fill in validated quality of life questionaires at all treatments.

To evaluate the effect of the treatment, all patients will be evaluated with standard CT scans prior to treatment and 3 and 9 months after the 4th treatment. Ga-68 DOTATOC PET will be performed at baseline and 6 and 12 months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients 18 years of age or more
* 2. NEN confirmed by histology
* 3. Clinical, PET/CT or CT proven progression despite standard treatment with somatostatin analogues, targeted therapy (Everolimus, sunitinib), chemotherapy (STZ/5-FU, temozolomide/capecitabine) OR intolerable side effects caused by these standard treatment OR unmanageable carcinoid symptoms
* 4. WHO/ ECOG Performance Status of 0-2
* 5. Life expectancy more than 6 months
* 6. Uptake higher than liver in primary tumor or metastases on Ga-DOTATOC PET/CT (Krenning 3 or 4), if the scan is more than 3 months old at inclusion time, a new scan should be done.
* 7. Adequate organ function as defined by:
* Adequate kidney function: Patient glomerular filtration rate >30 ml/min measured by Tc-DTPA clearance
* Adequate bone marrow function:

  * WBC ≥ 2.0 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hb ≥ 6 mmol/l (≥9.67 g/dL)
* 8. Willingness and ability to comply with scheduled visits for SPECT/CT scans, treatment plans, laboratory tests and other study procedures.

  9. Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

* 1. Tumor amenable to surgery and/or radiofrequency ablation
* 2. Patients who are unable to stay isolated for 24 hours
* 3. Previous PRRT
* 4. Female patients who are pregnant or lactating. Women who are of childbearing potential (defined as all women physiologically capable of becoming pregnant) have to practice an effective method of contraception/birth control. Fertile female patients have to take a urinary pregnancy test, to ensure that they are not pregnant, before they can enter the study. After entering the study, they have to use effective contraception during the study period and 6 months after. Effective contraception methods include:
* Use of oral, injected or implanted hormonal methods of contraception or
* Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Total abstinence or patient sterilization (male or female)
* 5. Male patients are not allowed to conceive pregnancy for 6 months after last treatment cycle
* 6. Known to be hypersensitive to any component of the Lu-177-DOTATOC
* 7. Patients with meningioma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months after LPLV
  Defined as time from randomization to documented disease progression or death by any cause, evaluated by CT, RECIST 1.1.

SECONDARY OUTCOMES:
Tumor dose | Through out the study efter each patient has completed treatment, up to 48 weeks
  Difference in tumor dose between dosimetry based and standard PRRT treatment groups and between patients in the dosimetry based treatment group over time.

OTHER OUTCOMES:
Kidney toxicity | At baseline and after 3, 6 and 12 months
  Measured by Tc-DTPA clearance
Kidney toxicity | At baseline and 3 months after the last treatment
  Measured by kidney fibrosis markers PRO-C6, PRO-C3, and C3M two groups
Bone marrow function, hemoglobin | Every second week in up to 64 weeks
  Measured by hemoglobin in the two groups
Bone marrow function, white blood cells | Every second week in up to 64 weeks
  Measured by white blood cells in the two groups
Bone marrow function, platelets | Every second week in up to 64 weeks
  Measured by platelets in the two groups
Subjective side effects | After every treatment, up to 48 weeks
  Evaluated by use of dedicated questionaire with score from 0-3
Quality of life score 1 | After every treatment, up to 48 weeks
  Evaluated by questionnaire EORTC QLQ-30 filled out at every treatment
Quality of life score 2 | After every treatment, up to 48 weeks
  Evaluated by questionnaire QLQ-GI.NET21. filled out at every treatment
Overall survival | 3 years after LPLV
  Registration of time for baseline to death

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, department of Nuclear medicine and PET centre, Aarhus, Palle Juul-Jensens Boulevard, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Franco M, Zanoni L, Fortunati E, Fanti S, Ambrosini V. Radionuclide Theranostics in Neuroendocrine Neoplasms: An Update. Curr Oncol Rep. 2024 May;26(5):538-550. doi: 10.1007/s11912-024-01526-5. Epub 2024 Apr 6. PMID 38581469